CLINICAL TRIAL: NCT04680208
Title: Reasons and Outcomes of Direct Admission of Surgical Patients to ICU: A Three Years Retrospective Study at University Hospital
Brief Title: Study of Direct Admission of Postoperative Patients to ICU
Status: Completed | Type: Observational
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Principal Investigator, Dr Jyoti Barud, Consultant Intensivist, Sultan Qaboos University
Other Study IDs: MREC#1937
Record Dates: First submitted 2020-12-07; First posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Postoperative Complications; Comorbidities and Coexisting Conditions
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Planned ICU admission: Cases who were planned for postoperative ICU admission at the time of preanesthetic check up
  Interventions: Procedure: Surgical procedure under anesthesia
- Unplanned ICU admission: Cases who got admitted to ICU postoperatively without anticipation
  Interventions: Procedure: Surgical procedure under anesthesia

INTERVENTIONS:
Procedure: Surgical procedure under anesthesia — Different varieties of surgical procedures done under anesthesia

SUMMARY:
Background: This study assessed perioperative factors associated with planned and unplanned postoperative ICU admission and evaluated the outcome of the two groups. There are limited researches evaluating these factors. Hence, it is important to do an audit that assesses the perioperative factors to help creating a criteria for postoperative ICU admissions.

Materials and methods: This retrospective study evaluated medical records of 68 patients above 18 years between January'2016- December'2018 that were admitted to ICU postoperatively in Sultan Qaboos University hospital in Oman. Both planned and unplanned admissions were assessed who underwent elective as well as emergency surgeries. Neurologic and cardiothoracic surgeries were excluded. Data collected included patient's demographics, social status like smoking, ASA physical status (American Society of Anesthesiologists), associated comorbidities, other perioperative factors and investigations, surgical and anesthesia details were recorded. The primary outcome studied was reasons of admission for planned versus unplanned postoperative ICU admissions. The secondary outcomes included mortality outcome and length of stay in ICU.

DETAILED DESCRIPTION:
There are 2 Levels of care available for patients who require high level of organ support and monitoring. First of them is the high dependency unit (HDU) where higher level organ support and monitoring is given (exception for mechanical ventilation) such as invasive blood pressure monitoring. Second one is the intensive care unit (ICU), which provides support for patients with multiple organ dysfunction that needs higher level of care which cannot be provided in the ward or the high dependency unit (HDU) and without this care the patient may not survive.

ICU admission post-operatively can be either in a planned or unplanned way. The complex interaction between associated comorbidities, anticipated complications intra-operatively and high American Society of Anesthesiologists (ASA) Physical Status are major factors in planning for ICU admission post-operatively. ASA physical status indicates patient's health status and has been accepted as a determinant of comorbidity and mortality. Unplanned ICU admissions can be due to unpredicted surgical or anesthetic intra-operative complications or poor assessment of perioperative factors. After surgery, some patients are admitted to ICU for further management and monitoring based on their underlying low functional status and co-morbidities. Out of these some patients may actually need ICU interventions and others may not. If an ICU bed is booked for unworthy patient, this may lead to unnecessary increased expenditure, wastage of valuable resources as well as deny the ICU services to potentially survivable and worthy critically ill patient.

This study aimed to assess perioperative factors associated with planned and unplanned admissions to find out the main reasons of admission to ICU at Sultan Qaboos University hospital (SQUH). This will help to lay guideline for guiding future admission to ICU for surgical patients in immediate postoperative period and help to reduce the unplanned admission.

Methods

This retrospective observational study traced all adult patients (above 18 years old) who underwent surgery and got admitted to ICU directly from operating theatre during the 3-year period: 2016-2018 at SQUH. These were segregated into planned and unplanned admissions. Required information was accessed using the hospital information system after receiving the ethical approval from Sultan Qaboos University Hospital Ethics and Research Committee (MREC#1937). Patients who were admitted to specialized ICU and those who underwent neurologic or cardiothoracic operations were excluded from this study since they are admitted postoperatively to ICU by default.

Patient's data that were collected included age, gender, social status like smoking, ASA physical status (American Society of Anesthesiologists), associated comorbidities such as diabetes, hypertension, ischemic heart disease, valvular heart disease, pulmonary diseases, chronic kidney disease and cirrhosis. Associated factors and investigations were collected like dehydration, hypoxia, hypercarbia, pH changes, pulmonary complications, fluid/electrolyte imbalance, temperature changes, random blood sugar, sepsis, coagulopathy, elevated WBC, low hemoglobin, hemodynamic instability, septic shock, hypovolemic shock, infection, blood loss more than 20%, hypotension and cardiac arrhythmia. Type, nature and duration of surgery, type of anesthesia and airway issues were recorded. Patients mortality outcome and length of stay in ICU were included as well.

Statistical methods: Statistical Package for the Social Sciences (SPSS) was used for patient's data analysis. Descriptive statistics were used to determine median, frequencies and percentages of the data and were presented in form of graphs and tables. For testing the significance between the way of ICU admission (planned/unplanned) and different variables, Chi-square and Fisher's exact test were used. To assess risk factors of mortality outcome and long ICU stay, odds ratio was used. P-value of 0.05 or less was considered to be significant.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over the age of 18 who underwent surgery and got admitted directly to ICU postoperatively

Exclusion Criteria:

* Patients who were admitted to specialized ICU ( cardiothoracic and neurosurgery ) or to the ward and then ICU
* Pediatric patients

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (above 18 years old) who underwent surgery and got admitted to ICU directly from operating theatre
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Reasons of admission for postoperative ICU patients. | 1-2 days
  Study of main reasons of ICU admissions directly from operating room. The reasons like type of surgery, ASA grading, preoperative functional status, co-morbidities: diabetes, hypertension, ischemic heart disease etc, intraoperative events like hemodynamic instability/shock, respiratory compromise, prolonged duration of surgery and other anesthesia complications will be studied as reasons of admission for planned versus unplanned ICU admissions for postoperative patients.

SECONDARY OUTCOMES:
ICU length of stay | 1-30 days
Mortality | 1-45 days
  Postoperative mortality

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti Burad, M.D E.D.I.C, Principal Investigator — Sultan Qaboos University Hospital; Batool Al Ajmi, Student, Principal Investigator — Sultan Qaboos University Hospital
Locations (1):
- Sultan Qaboos University Hospital,, Muscat, Oman

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Meziane M, El Jaouhari SD, ElKoundi A, Bensghir M, Baba H, Ahtil R, Aboulaala K, Balkhi H, Haimeur C. Unplanned Intensive Care Unit Admission following Elective Surgical Adverse Events: Incidence, Patient Characteristics, Preventability, and Outcome. Indian J Crit Care Med. 2017 Mar;21(3):127-130. doi: 10.4103/ijccm.IJCCM_428_16. PMID 28400682
- [Background] Pearse RM, Harrison DA, James P, Watson D, Hinds C, Rhodes A, Grounds RM, Bennett ED. Identification and characterisation of the high-risk surgical population in the United Kingdom. Crit Care. 2006;10(3):R81. doi: 10.1186/cc4928. Epub 2006 Jun 2. PMID 16749940
- [Background] Smith G, Nielsen M. ABC of intensive care. Criteria for admission. BMJ. 1999 Jun 5;318(7197):1544-7. doi: 10.1136/bmj.318.7197.1544. No abstract available. PMID 10356016
- [Background] Sobol JB, Wunsch H. Triage of high-risk surgical patients for intensive care. Crit Care. 2011;15(2):217. doi: 10.1186/cc9999. Epub 2011 Mar 22. No abstract available. PMID 21457500
- [Result] Patel SK, Kacheriwala SM, Duttaroy DD. Audit of Postoperative Surgical Intensive Care Unit Admissions. Indian J Crit Care Med. 2018 Jan;22(1):10-15. doi: 10.4103/ijccm.IJCCM_387_17. PMID 29422726